CLINICAL TRIAL: NCT03556657
Title: MUSic Therapy to Improve Quality Of Life in Sickle Cell Disease (MUSIQOLS): A Pilot Study
Brief Title: MUSic Therapy to Improve Quality Of Life in Sickle Cell Disease (MUSIQOLS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Kulas Foundation (Other)
Responsible Party: Principal Investigator, Samuel Rodgers-Melnick, Music Therapist, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20180101
Record Dates: First submitted 2018-05-22; First posted 2018-06-14 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Sickle Cell Disease; Chronic Pain
Keywords: Music Therapy; Sickle Cell Disease; Quality of Life; Chronic Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Chronic Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy Group (Experimental): Patient receives 6 sessions of music therapy with a board-certified music therapist. Patient will learn various music interventions for pain management that he/she will utilize at home.
  Interventions: Other: Music Therapy
- Wait-List Control Group (No Intervention): Patient receives standard care alone. Patient will receive music therapy sessions following completion of the post-test.

INTERVENTIONS:
Other: Music Therapy — Patient receives 6 sessions of music therapy with a board-certified music therapist. Patient will learn various music interventions for pain management that he/she will utilize at home.
  Arms: Music Therapy Group

SUMMARY:
The purpose of this pilot study is to investigate the effects of a 6-session music therapy protocol on the pain, mood, quality of life, coping skills, and self-efficacy of adult patients with sickle cell disease (SCD) as compared to adult patients with SCD who receive standard care alone. The investigators will also determine the feasibility (delivery, acceptability, and usefulness) of the music therapy intervention for pain management and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older
* Subject has a SCD diagnosis
* Subject fits chronic pain criteria in SCD
* Subject has a working email address
* Subject has access to a mobile device with email and internet capabilities
* Subject is able to speak and understand English
* Subject has attended at least 50% of his/her scheduled outpatient visits to the Adult SCD Clinic in the last 12 months

Exclusion Criteria:

* Subject has a significant visual impairment that has not been corrected
* Subject has a significant hearing impairment that has not been corrected
* Subject has a significant cognitive impairment that would prevent subject from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 4a | Pre-test at baseline and post-test at 10 weeks
  Physical function (4 questions)
Change from baseline in Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) | Pre-test at baseline and post-test at 10 weeks
  A patient-reported outcome measurement system that addresses the physical, social, and emotional impact of SCD. ASCQ-Me scores are calculated in the direction of overall health, with higher ASCQ-Me scores indicating better health.
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety Short Form 4a | Pre-test at baseline and post-test at 10 weeks
  Anxiety (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression - Short Form 4a | Pre-test at baseline and post-test at 10 weeks
  Depression (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue - Short Form 4a | Pre-test at baseline and post-test at 10 weeks
  Fatigue (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities - Short Form 4a | Pre-test at baseline and post-test at 10 weeks
  Ability to participate in social roles and activities (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference - Short Form 4a | Pre-test at baseline and post-test at 10 weeks
  Pain interference (4 questions)

SECONDARY OUTCOMES:
Change from baseline in Sickle Cell Self-Efficacy Scale (SCSES) | Pre-test at baseline and post-test at 10 weeks
  A nine-item Likert scale originally developed for adults with SCD to assess patients' beliefs in their ability to manage their own SCD.
Change from baseline in Coping Skills Questionnaire - Sickle Cell Disease (CSQ-SCD) | Pre-test at baseline and post-test at 10 weeks
  80-item questionnaire that assesses coping strategies relevant to SCD
Electronic Sickle Cell Disease Pain Diary | Daily entries for 2 weeks at baseline and daily entries for 2 weeks post-intervention
  A multidimensional pain diary assessing daily pain intensity, location, description, cause, and interference with daily activities
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance - Short Form 4a | Pre-test at baseline and post-test at 10 weeks
  Sleep disturbance (4 questions)

OTHER OUTCOMES:
Semi-structured interview | At post-test at 10 weeks
  Interview questions will focus on the patient's current pain, his/her experience of the music therapy sessions, and whether anything could have been done differently to improve the music therapy sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel N Rodgers-Melnick, MT-BC, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Seidman Cancer Center, Cleveland, Ohio, United States